CLINICAL TRIAL: NCT01096290
Title: Comparison of Lubiprostone and Placebo for the Relief of Constipation From Constipating Medications
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Number of needed participants could not be obtained
Sponsor: University of South Alabama (Other)
Collaborators: Takeda (Industry); Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-250
Record Dates: First submitted 2010-03-22; First posted 2010-03-31 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Constipation
Keywords: constipation; lubiprostone; healthy volunteers
MeSH Terms: conditions — Constipation | interventions — Lubiprostone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lubiprostone 24mcg BID for 30 days (Experimental): Active medication
  Interventions: Drug: lubiprostone
- Placebo (Placebo Comparator): Placebo, matched, blinded
  Interventions: Drug: Matched placebo

INTERVENTIONS:
Drug: lubiprostone — 24mcg BID, capsule, oral 30days
  Other Names: Amitiza
  Arms: Lubiprostone 24mcg BID for 30 days
Drug: Matched placebo — Twice daily for 30days, oral
  Other Names: Placebo, sugar pill
  Arms: Placebo

SUMMARY:
Constipation from medications is a serious and common condition. Lubiprostone has properties that make it a candidate drug. One hundred volunteers with constipation who are taking medications known to cause constipation will be randomized to take lubiprostone or placebo for 28 days. Therapeutic outcome will be evaluated by investigator and study subject assessment.

DETAILED DESCRIPTION:
Lubiprostone is a novel chloride channel activator that increases intestinal fluid secretion and motility. It is FDA approved and indicated for treatment of chronic idiopathic constipation and recently, constipation-predominant irritable bowel syndrome.

The Physicians Desk Reference lists over 90 Brand medications with reported incidence associated with constipation over 3%. Little data are available about treatment responses. A recent publication by our group reported treatment success for medication constipation using polyethylene glycol. Since ongoing studies are addressing the role of lubiprostone in opioid constipation, this work will be enrolling medication constipation study subjects not using opioids.

In this study, patients who meet diagnostic criteria for constipation will be randomized to receive 28 days of treatment with lubiprostone 24mcg twice a day. Data will be collected to evaluate therapeutic outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female outpatient age 19 or older.
* Patients meet International Congress of Gastroenterology (ROME III) clinical criteria for constipation*:

  1. Must include two or more of the following:

     1. Straining in > 1/4 defecations;
     2. Lumpy or hard stools > 1/4 defecations;
     3. Sensation of incomplete evacuation in 1/4 defecations;
     4. Sensation of anorectal obstruction/blockage in > 1/4 defecations;
     5. <3 defecations/week.
  2. Loose stools are rarely present without the use of laxatives.
  3. There are insufficient criteria for irritable bowel syndrome. *Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.
* Use of one or more of listed medications known to cause constipation.
* If female and of childbearing potential, patient must be surgically sterilized or using oral contraceptives, depot contraceptives, intrauterine device, or testifies that she is monogamous with a vasectomized partner, or practices abstinence and will continue to do so during the duration of study. Mandatory compliance is required. Serum pregnancy tests will be performed at screening and during needed follow-up. Negative results will be received before inclusion and administration of first study dose. If pregnancy occurs during the trial, the investigator is notified immediately resulting in prompt discontinuation.
* Study subjects must not have received lubiprostone for more than 72 hours.
* Written informed consent.

Exclusion Criteria:

* Known or suspected obstruction, gastric retention, ileus, perforation, fecal impaction or inflammatory bowel disease.
* Severe diarrhea.
* Prior small bowel or colonic resection or colostomy.
* Weight < 80 lbs.
* If the patient has constipation that according to the investigator's clinical judgment is not the result of constipating medications but is suffering from a secondary cause including but limited to factors that are dietary, neurologic, congenital, diabetic or hypothyroid.
* Positive stool hemoccult (Can be included if colonoscopic evaluation is subsequently negative).
* Significant cardiac, renal or hepatic insufficiency.
* Pregnant or expecting to become pregnant within 120 days of study enrollment.
* Lactating or breast feeding.
* Subjects using opioid medications.
* Subjects who in the opinion of the investigator would be unable to comply adequately with the study plan.
* Use of investigational drugs in the last 30 days.
* Patients with known allergy to lubiprostone.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A DiPalma, M.D., Principal Investigator — University of South Alabama College of Medicine
Locations (1):
- USA Pavilion at Infirmary West, Mobile, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lubiprostone 24mcg BID for 30 Days | Placebo
Started | 9 | 14
Completed | 9 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone 24mcg BID for 30 Days | Placebo | Total
Number analyzed (Participants) | 9 | 14 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 20
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Relief of Constipation Defined by Modified ROME Criteria
Description: Subjects will report symptoms by questionnaire
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lubiprostone 24mcg BID for 30 Days | Placebo
Number analyzed (Participants) | 9 | 14
Participants | 7 | 7

2. Secondary Outcome: Frequency
Description: Subjects will report stool frequency by questionnaire
Time Frame: 30 days
Population: Data was not collected for this Outcome Measure
Arm/Group | Lubiprostone 24mcg BID for 30 Days | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From screening visit 1 to Follow-up Day 56
Arm/Group | Lubiprostone 24mcg BID for 30 Days | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/14
Other Adverse Events (participants affected / at risk) | 0/9 | 0/14

LIMITATIONS AND CAVEATS:
100 participants were needed to obtain statistical power. Only 23 participants were enrolled. Therefore, data analysis was not completed since a success rate could not be adequately demonstrated on such a small sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes